CLINICAL TRIAL: NCT01223378
Title: A Randomized, Multicenter, Single-Masked, Parallel-Group Dose Finding Study Comparing the Safety and Efficacy of BOL-303259-X to Latanoprost in Subjects With Open Angle Glaucoma or Ocular Hypertension
Brief Title: Study Comparing the Safety and Efficacy of BOL-303259-X to Latanoprost in Subjects With Glaucoma or Ocular Hypertension
Acronym: Voyager
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 659
Record Dates: First submitted 2010-10-11; First posted 2010-10-19 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Intraocular Pressure
MeSH Terms: interventions — BOL 303259-X; Latanoprost

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BOL-303259-X (Experimental): ophthalmic solution
  Interventions: Drug: BOL-303259-X
- Latanoprost (Active Comparator): ophthalmic solution
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: BOL-303259-X — ophthalmic solution, various concentrations, once daily (QD) 28 days
  Other Names: latanoprostene bunod
  Arms: BOL-303259-X
Drug: Latanoprost — 0.005% ophthalmic solution, QD 28 days
  Other Names: Xalatan
  Arms: Latanoprost

SUMMARY:
The objective of this clinical investigation is to determine the most effective drug concentration(s) of BOL-303259-X in the reduction of IOP in order to support further clinical development of an appropriate dose with regard to efficacy, and ocular and systemic safety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of open angle glaucoma (OAG) or ocular hypertension (OH) in one or both eyes.
* IOP requirements at Visit 3, A mean/median IOP ≥ 26 mmHg at a minimum of 1 time point, ≥ 24 mmHg at a minimum of 1 time point, and ≥ 22 mmHg at 1 time point in the same eye, and Mean/median IOP ≤ 32 mmHg in both eyes at all 3 measurement time points.
* Subjects with best-corrected visual acuity (BCVA), using Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol, of +0.7 logMAR units (Snellen equivalent ~20/100) or better in either eye.

Exclusion Criteria:

* Subjects with a known hypersensitivity or contraindications to latanoprost or any of the ingredients in the study drugs.
* Subjects with known contraindications to nitric oxide (NO) treatment.
* Subjects whose central corneal thickness was greater than 600um in either eye.
* Subjects with any condition that prevented reliable applanation tonometry in either eye.
* Subjects with advanced glaucoma and subjects with a cup/disc ratio greater than 0.8 or a history of split fixation, or a field loss threatening fixation in either eye.
* Subjects with previous or active corneal disease.
* Subjects with a history of severe dry eye.
* Subjects with monophthalmia.
* Subjects with optic disc hemorrhage.
* Subjects with a history of central retinal vein and artery occlusion.
* Subjects with a history of macular edema.
* Subjects with any intraocular infection, inflammation, or laser surgery within the previous 6 months from Visit 1 (Screening).
* Subjects who had incisional ocular surgery or severe trauma within the previous 6 months from Visit 1 (Screening).
* Subjects with very narrow angles (3 quadrants with less than Grade 2 according to Shaffer's anterior chamber angle grading system) and subjects with angle closure, congenital and secondary glaucoma, and subjects with history of angle closure in either eye.
* Subjects with a diagnosis of a clinically significant or progressive retinal disease in either eye.
* Subjects who were expected to require treatment with ocular or systemic corticosteroids.
* Subjects who were in need of any other topical or systemic treatment of OAG or OHT.
* Subjects with an anticipated need to initiate or modify medication (systemic or topical) that was known to affect IOP during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2011-12-20 (Actual); Study Completion 2012-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Ozden, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Inc, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weinreb RN, Ong T, Scassellati Sforzolini B, Vittitow JL, Singh K, Kaufman PL; VOYAGER study group. A randomised, controlled comparison of latanoprostene bunod and latanoprost 0.005% in the treatment of ocular hypertension and open angle glaucoma: the VOYAGER study. Br J Ophthalmol. 2015 Jun;99(6):738-45. doi: 10.1136/bjophthalmol-2014-305908. Epub 2014 Dec 8. PMID 25488946

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled on 13 Dec 2010, Last subject exited on 20 Dec 2011. This study was conducted at 23 clinical sites. US [15 sites], Bulgaria [3 sites], Poland [3 sites], and Czech Republic [2 sites]).
Pre-assignment Details: Subjects who were currently under treatment with an IOP-lowering medication at Visit 1 were required to discontinue the IOP medication during the washout period (minimum of 28 days) between Visit 1 and Visit 3.
Groups:
- BOL-303259-X 0.006%: ophthalmic solution
  Experimental: BOL-303259-X: ophthalmic solution, 0.006%, once daily (QD) 28 days
- BOL-303259-X 0.012%: ophthalmic solution
  Experimental: BOL-303259-X: ophthalmic solution, 0.012%, once daily (QD) 28 days
- BOL-303259-X 0.024%: ophthalmic solution
  Experimental: BOL-303259-X: ophthalmic solution, 0.024%, once daily (QD) 28 days
- BOL-303259-X 0.040%: ophthalmic solution
  Experimental: BOL-303259-X: ophthalmic solution, 0.040%, once daily (QD) 28 days
Period: Overall Study
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Started | 82 | 85 | 83 | 81 | 82
Completed | 76 | 81 | 80 | 80 | 79
Not Completed | 6 | 4 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost | Total
Number analyzed (Participants) | 82 | 85 | 83 | 81 | 82 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (11.39) | 61.6 (9.58) | 60.8 (11.47) | 60.3 (12.89) | 61.2 (11.92) | 61.0 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 46 | 57 | 43 | 53 | 255
  Male | 26 | 39 | 26 | 38 | 29 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 8 | 6 | 11 | 32
  Not Hispanic or Latino | 77 | 83 | 75 | 75 | 71 | 381
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 21 | 23 | 21 | 23 | 16 | 104
  White | 61 | 61 | 62 | 56 | 66 | 306
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Diurnal IOP at Visit 6 (Day 28)
Description: Determine the most effective drug concentration(s) of BOL-303259-X in the reduction of intraocular pressure (IOP) and compared to latanoprost
Time Frame: Baseline and Visit 6 (Day 28)
Population: Intent-to-treat population, observed data (study eye)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Number analyzed (Participants) | 81 | 83 | 83 | 80 | 80
mm Hg | -7.829 (2.823) | -8.295 (2.864) | -8.952 (3.337) | -8.894 (2.666) | -7.800 (2.834)

2. Secondary Outcome: Change in Mean Diurnal IOP at Visits 4,5, and 7
Description: as for outcome 1
Time Frame: Baseline and Visit 4 (Day 7), Visit 5 (day 14), and Visit 7 (Day 29)
Population: Intent-to-treat population, observed data (study eye)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Number analyzed (Participants) | 79 | 82 | 81 | 80 | 80
mm Hg
  Visit 4 (Day 7) | -6.850 (2.768) | -7.707 (3.192) | -8.230 (3.286) | -8.456 (2.892) | -7.325 (2.699)
  Visit 5 (Day 14): number analyzed (Participants) | 76 | 80 | 80 | 80 | 79
  Visit 5 (Day 14) | -7.607 (2.204) | -7.934 (3.065) | -8.859 (3.300) | -8.606 (2.878) | -7.719 (3.035)
  Visit 7 (Day 29): number analyzed (Participants) | 76 | 81 | 80 | 80 | 79
  Visit 7 (Day 29) | -6.188 (2.782) | -6.202 (3.001) | -7.177 (3.615) | -6.846 (3.135) | -6.276 (2.941)

3. Secondary Outcome: IOP </=18mm Hg
Description: Determine the number of subjects with mean diurnal IOP </=18 mm Hg with BOL-303259-X versus latanoprost ophthalmic solution
Time Frame: Visit 4 (Day 7), Visit 5 (day 14), Visit 6 (Day 28) and Visit 7 (Day 29)
Population: Intent-to-treat population, observed data (study eye)
Measure: Count of Participants; unit: Participants
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Number analyzed (Participants) | 82 | 85 | 83 | 81 | 82
Participants
  Visit 4 (Day 7): number analyzed (Participants) | 79 | 82 | 81 | 80 | 80
  Visit 4 (Day 7) | 30 | 37 | 47 | 46 | 29
  Visit 5 (Day 14): number analyzed (Participants) | 76 | 80 | 80 | 80 | 79
  Visit 5 (Day 14) | 34 | 42 | 52 | 45 | 39
  Visit 6 (Day 28): number analyzed (Participants) | 81 | 83 | 83 | 80 | 80
  Visit 6 (Day 28) | 41 | 44 | 57 | 51 | 38
  Visit 7 (Day 29): number analyzed (Participants) | 76 | 81 | 80 | 80 | 79
  Visit 7 (Day 29) | 25 | 24 | 37 | 25 | 23

4. Secondary Outcome: Change in IOP at Specified Time Points (8 AM, 12 PM, 4 PM) at Visit 6 (Day 28)
Description: The change in the observed mean study eye IOP from baseline (Visit 3, Day 1) at specified time points (8 AM, 12 PM, 4 PM) at Visit 6 (Day 28)
Time Frame: baseline and Visit 6 (Day 28)
Population: Intent to treat, data as observed (study eye)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Number analyzed (Participants) | 82 | 85 | 83 | 81 | 82
mm Hg
  Change from Baseline (8 am): number analyzed (Participants) | 81 | 83 | 83 | 80 | 80
  Change from Baseline (8 am) | -8.42 (3.69) | -8.91 (3.24) | -9.46 (4.01) | -9.61 (2.95) | -8.76 (3.24)
  Change from Baseline (12 pm): number analyzed (Participants) | 79 | 83 | 82 | 80 | 79
  Change from Baseline (12 pm) | -7.82 (3.34) | -8.33 (3.35) | -8.98 (3.50) | -8.60 (3.23) | -7.63 (3.55)
  Change from Baseline (4 pm): number analyzed (Participants) | 79 | 83 | 82 | 80 | 79
  Change from Baseline (4 pm) | -7.23 (2.97) | -7.65 (3.37) | -8.59 (3.54) | -8.47 (3.28) | -6.99 (3.52)

5. Secondary Outcome: Change in IOP at Specified Time Points (8 AM, 12 PM, 4 PM) at Visits 4, 5, and 7 (Days 7, 14, and 29)
Description: The change in the observed mean study eye IOP from baseline (Visit 3, Day 1) at specified time points (points 8 AM, 12 PM, and 4 PM) at Visits 4, 5, and 7 (Days 7, 14, and 29)
Time Frame: baseline and Visits 4, 5 and 7 (Days 7, 14, and 29)
Population: Intent-to-treat, observed data (study eye)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
Number analyzed (Participants) | 79 | 82 | 81 | 80 | 80
mm Hg
  Visit 4 (Day 7) (8 am) | -7.203 (3.634) | -8.396 (3.935) | -8.667 (3.827) | -8.869 (3.384) | -8.125 (2.826)
  Visit 4 (Day 7) (12 pm) | -6.665 (3.046) | -7.823 (3.409) | -8.247 (3.643) | -8.219 (3.338) | -7.200 (3.386)
  Visit 4 (Day 7) (4 pm) | -6.684 (3.246) | -6.902 (3.371) | -7.778 (3.479) | -8.281 (3.172) | -6.650 (3.312)
  Visit 5 (Day 14) (8 am): number analyzed (Participants) | 76 | 80 | 80 | 80 | 79
  Visit 5 (Day 14) (8 am) | -8.270 (3.399) | -8.538 (3.518) | -9.569 (3.597) | -9.006 (3.031) | -8.519 (3.444)
  Visit 5 (Day 14) (12 pm): number analyzed (Participants) | 76 | 80 | 80 | 80 | 79
  Visit 5 (Day 14) (12 pm) | -7.500 (2.653) | -8.381 (3.518) | -8.700 (3.579) | -8.556 (3.529) | -7.519 (3.437)
  Visit 5 (Day 14) (4 pm): number analyzed (Participants) | 76 | 79 | 79 | 80 | 79
  Visit 5 (Day 14) (4 pm) | -7.053 (2.519) | -6.905 (3.354) | -8.310 (3.667) | -8.256 (3.410) | -7.120 (3.744)
  Visit 7 (Day 29) (8 am): number analyzed (Participants) | 76 | 81 | 80 | 80 | 79
  Visit 7 (Day 29) (8 am) | -6.969 (3.245) | -6.796 (3.379) | -7.675 (4.198) | -7.406 (3.26) | -7.006 (3.131)
  Visit 7 (Day 29) (12 pm): number analyzed (Participants) | 76 | 81 | 80 | 79 | 79
  Visit 7 (Day 29) (12 pm) | -6.039 (3.591) | -6.235 (3.626) | -7.119 (3.791) | -6.791 (3.246) | -6.108 (3.228)
  Visit 7 (Day 29) (4 pm): number analyzed (Participants) | 73 | 81 | 80 | 78 | 79
  Visit 7 (Day 29) (4 pm) | -5.575 (3.464) | -5.574 (3.615) | -6.738 (3.769) | -6.090 (4.142) | -5.715 (3.514)

ADVERSE EVENTS:
Time Frame: The period of observation for collection of AEs extended from the time the subject gave informed consent until the last study visit (Visit 7).
Description: The safety population included one less subject in the BOL-303259-X 0.012% group than the ITT population. Hence the safety population included 412 subjects in total whereas the ITT population included 413 in total.
Arm/Group | BOL-303259-X 0.006% | BOL-303259-X 0.012% | BOL-303259-X 0.024% | BOL-303259-X 0.040% | Latanoprost
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/84 | 0/83 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/82 | 0/84 | 0/83 | 0/81 | 2/82
Other Adverse Events (participants affected / at risk) | 20/82 | 18/84 | 20/83 | 23/81 | 10/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOL-303259-X 0.006% (N=82) | BOL-303259-X 0.012% (N=84) | BOL-303259-X 0.024% (N=83) | BOL-303259-X 0.040% (N=81) | Latanoprost (N=82)
Gastric Ulcer Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Bleeding gastric ulcer
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Acute myocardial infarction
Gastrointestinal Hemorrage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Gastrointestinal bleed
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Gastric Ulcer
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOL-303259-X 0.006% (N=82) | BOL-303259-X 0.012% (N=84) | BOL-303259-X 0.024% (N=83) | BOL-303259-X 0.040% (N=81) | Latanoprost (N=82)
Ocular Hyperemia (Eye disorders) | 1 (1) | 5 (5) | 2 (2) | 4 (4) | 7 (7)
Conjunctival Hyperemia (Eye disorders) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 0 (0)
Eye Irritation (Eye disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 0 (0)
Instillation Site Pain (General disorders) | 12 (12) | 14 (14) | 10 (10) | 14 (14) | 5 (5)
Punctate Keratitis (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal Sensation in the Eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Keratopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Follicles (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Lid Edema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Growth of Eyelashes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation Site Erythema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Instillation Site Lacrimation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Instillation Site Pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Instillation Site Reaction (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Instillation Site Discomfort (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Instillation Site Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine with Aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No